CLINICAL TRIAL: NCT03394027
Title: A Phase 2 Study of ONC201 in Recurrent/Refractory Metastatic Breast Cancer and Advanced Endometrial Carcinoma
Brief Title: ONC201 in Recurrent/Refractory Metastatic Breast Cancer and Advanced Endometrial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stanley Lipkowitz, MD, PhD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180034; 18-C-0034
Record Dates: First submitted 2018-01-05; First posted 2018-01-09 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-07

CONDITIONS: Triple Negative Breast Cancer; Endometrial Cancer; Hormone Receptor Positive, HER2 Negative Breast Cancer
Keywords: Imipridones; TNBC; Metastatic; Male Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Endometrial Neoplasms; Neoplasm Metastasis; Breast Neoplasms, Male | interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1-ONC201 in Recurrent/Refractory Metastatic Breast Cancer and Advanced Endometrial Carcinoma (Experimental): Single arm divided in three cohorts, each cohort with a different type of metastatic disease: estrogen receptor (ER) + breast cancer, triple negative breast cancer, and endometrial cancer
  Interventions: Drug: ONC201

INTERVENTIONS:
Drug: ONC201 — 625 mg by mouth every 7 days; each cycle = 28 days. Patients will receive ONC201 as long as they derive clinical benefit or toxicity becomes impeditive.

SUMMARY:
Background:

The new drug ONC201 have been shown to kill breast cancer and endometrial cancer cells in the laboratory. The exact mechanism of action is not completely clear yet, but the ONC201 destroys the mitochondria inside the cells. Blocking mitochondrial activity may kill tumor cells, which would shrink tumors. Researchers want to see if ONC201 helps shrink tumors of certain breast or endometrial cancers and if that effect is maintained.

Objective:

To see if ONC201 shrinks tumors with a lasting effect.

Eligibility:

Adults ages 18 and older who have metastatic breast cancer (hormone-positive or triple-negative) or metastatic endometrial cancers.

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Heart, blood, and urine tests
* Computed tomography (CT) and bone scans
* Review of medical report and tumor sample
* Participants will have a tumor biopsy before starting treatment and after 5 weeks taking the study drug. A scan or ultrasound may be used to guide the biopsy. Patients will receive local anesthetic and a needle will remove a small piece of tumor.
* The study will be done in 28-day cycles. Every day 1 of each cycle participants will repeat most screening tests, will be seen by the physician and receive a supply of the study drug.
* Participants will take the study drug by mouth once every 7 days. They will keep a diary of when they take the drug and any side effects. During cycle 1, participants will get weekly calls to discuss their health and symptoms. Images will be repeated every 2 cycles to evaluate response to the treatment.

DETAILED DESCRIPTION:
Background:

* Advanced breast cancer and endometrial cancer have limited treatment options. Current treatments provide a modest improvement in progression free survival, but no treatments improve survival.
* ONC201 is the founding member of a novel class of anticancer drugs called imipridones. The exact mechanism of ONC201 is unknown at this time, but preclinical data suggests that it causes global downregulation of mitochondrial genes leading to mitochondrial damage and ultimately non-apoptotic cell death.
* Preclinical studies have demonstrated that ONC201 selectively kills various cancer cells, including breast cancer cells (hormone-receptor positive cell lines, human epidermal growth factor receptor 2 (HER2+) cell line as well as triple negative breast cancer cell lines) and endometrial cancer cells, while having little effect on normal cells.
* An on-going phase I study of ONC201 has demonstrated clinical benefit in some solid tumors, including endometrial cancer.

Objectives:

* Cohort 1: To determine the progression free survival (PFS) at 8 months of ONC201 in metastatic hormone receptor positive breast cancer (HR+BC)
* Cohort 2: To determine the overall response rate (ORR) of ONC201 in metastatic triple negative breast cancer (TNBC)
* Cohort 3: To determine the overall response rate (ORR) of ONC201 in advanced endometrial cancer (EC)

Eligibility:

Selected Inclusion Criteria

* Histologically confirmed metastatic breast cancer or endometrial cancer with appropriate immunohistochemistry (IHC) testing and confirmation of HER2 non-amplification required for the breast cancer cohorts (cohorts 1 and 2)
* Age 18 years or older
* Female and male breast cancer patients are eligible for the breast cancer cohorts
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Measurable metastatic disease with greater than or equal to 1 biopsiable lesion with willingness to undergo a biopsy
* Cohort 1 Hormone receptor + breast cancer (HR+BC) requires prior treatment with greater than or equal to 2 lines of hormonal treatment. No prior treatment required for cohorts 2/3 (TNBC and EC).
* Adequate hematopoietic, hepatic and renal function

Selected Exclusion Criteria

* Patients who have received chemotherapy in the previous 3 weeks (6 weeks for nitrosoureas or mitomycin); other investigational agents within 3 weeks or a programmed cell death protein 1 (PD1)/programmed death-ligand 1 (PDL1) agent within 4 weeks prior to first dose of study treatment.
* Radiotherapy less than or equal to 4 weeks before first dose of study treatment.
* Symptomatic central nervous system (CNS) metastases. Asymptomatic or brain metastases treated greater than 4 weeks from first dose of study treatment are allowed.
* History of invasive malignancy less than or equal to 3 years
* Known history of cardiac arrhythmias including uncontrolled atrial fibrillation, tachyarrhythmias or bradycardia.
* History of congestive heart failure (CHF), or myocardial infarction (MI) or stroke in the previous 3 months will be excluded.
* Started denosumab or bisphosphonate therapy within 28 days prior to Cycle 1 Day 1
* Human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C infection

Design:

* This is a phase II single arm study of ONC201 divided in three cohorts, each cohort with different type of metastatic, advanced disease:
* Cohort 1: HR+ breast cancer (male and female)
* Cohort 2: Triple negative breast cancer (male and female)
* Cohort 3: Endometrial cancer (female only)
* All patients will receive ONC201 at the recommended phase 2 dose (RP2D) of 625mg by mouth every 7 days with each cycle being 28 days long. Patients will receive ONC201 as long as they derive clinical benefit or toxicity becomes impeditive
* Patients will be evaluated for toxicity every 4 weeks by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and for response every two cycles (8 weeks) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

ELIGIBILITY:
* INCLUSION CRITERIA FOR COHORT 1: HORMONE RECEPTOR POSITIVE BREAST CANCER:
* Patients must have histologically confirmed persistent or recurrent invasive metastatic hormone receptor positive, human epidermal growth factor receptor 2 (HER2) normal breast cancer for which standard curative measures do not exist or are no longer effective. Hormone receptor positive is defined as estrogen receptor (ER) positive greater than or equal to 10% by immunohistochemistry (IHC) and/or progesterone receptor (PR) positive greater than or equal to 10% by IHC.HER2 will be considered negative per American Society of Clinical Oncology (ASCO)-College of American Pathologists (CAP) guidelines (HER2 test result as negative if a single test (or both tests) performed show: 1) IHC 1+ as defined by incomplete membrane staining that is faint/barely perceptible and within >10% of the invasive tumor cells; 2) IHC 0 as defined by no staining observed or membrane staining that is incomplete and is faint/barely perceptible and within less than or equal to 10% of the invasive tumor cells; or 3) ISH negative based on: a) Single-probe average HER2 copy number <4.0 signals/cell or b) Dualprobe HER2/ chromosome enumeration probe 17 (CEP17) ratio <2.0 with an average HER2 copy number <4.0 signals/cell)and HER2 testing must have been performed in a laboratory accredited by the College of American Pathologists (CAP) or another accrediting entity.
* Patients must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Patients must have at least one lesion deemed safe to biopsy and be willing to undergo mandatory biopsies.
* Hormone receptor + breast cancer (HR+BC) patients must have received prior treatment with at least 2 lines of hormonal treatment (Selective estrogen receptor modulators (SERM), aromatase inhibitor (AI), or fulvestrant) and deemed ineligible for further hormonal therapy. Patients may have received prior chemotherapy and there is no limit to the number of prior chemotherapy.
* Age greater than or equal to18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate renal function, defined as serum creatinine less than or equal to 1.5 X upper limit of normal (ULN), or measured creatinine clearance greater than or equal to 60 mL/min/1.
* Adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels less than or equal to 3 X ULN and total bilirubin < 1.5 X ULN, unless known diagnosis of Gilbert's syndrome, where bilirubin less than or equal to 5 mg/dL will be permitted. Gilbert's syndrome will be defined as elevated unconjugated bilirubin, with conjugated (direct) bilirubin within the normal range and less than 20% of the total. Total bilirubin will be permitted up to 5 mg/dL, if patients have historical readings consistent with the definition of Gilbert's syndrome prior to entering study.
* Adequate bone marrow function, defined as absolute neutrophil (ANC) greater than or equal to 1,500/mm^3 (greater than or equal to 1.5 X10^6/L), platelet count greater than or equal to 75,000/mm^3 (greater than or equal to 75 X10^6/L), and hemoglobin greater than or equal to 9 mg/dL (transfusion to obtain hemoglobin greater than or equal to 9 mg/dL within 24 hours prior to dosing is allowed).
* Patients must be able to swallow oral medications (capsules) without chewing, breaking, crushing, opening or otherwise altering the product formulation.
* The effects of ONC201 on the developing human fetus are unknown. For this reason and because imipridone agents are known to be teratogenic, female patients must either be of non-reproductive potential (i.e., post-menopausal by history: greater than or equal to 60 years old and no menses for greater than or equal to 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry and agree to use contraception or abstinence during the study and for and for at least 4 weeks after the final dose of any study-related medications. Male patients must use at least two forms of contraception during the study and for at least 4 weeks after the final dose of any study-related medications or have a partner who is not of reproductive potential.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA FOR COHORT 1: HORMONE RECEPTOR POSITIVE BREAST CANCER:

* Patients who have received chemotherapy in the previous 3 weeks (6 weeks for nitrosoureas or mitomycin); other investigational agents within 3 weeks or a programmed cell death protein 1 (PD1)/programmed death-ligand 1 (PDL1) agent within 4 weeks prior to first dose of study enrollment.
* Patients who have undergone radiotherapy within 4 weeks of first dose of study treatment.
* Patients with a history of another invasive malignancy within the last 3 years.
* Patients with symptomatic brain metastases or leptomeningeal involvement. Patients with asymptomatic or brain metastases that have been treated with radiation at least 4 weeks prior to first dose of study treatment are allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to imipridones or other agents used in study.
* Patients with a mean corrected Q wave T wave (QT) interval by Fridericia (QTcF) interval of > 500 msec or receiving therapeutic agents known to prolong the QT interval
* Known history of cardiac arrhythmias including uncontrolled atrial fibrillation, tachyarrhythmias or bradycardia, history of congestive heart failure, or myocardial infarction or stroke in the previous 3 months will be excluded.
* Known history of gastrointestinal illnesses that would preclude the absorption of ONC201, which is an oral agent.
* Patients with bone metastases who have initiated denosumab or bisphosphonate therapy within 28 days prior to Cycle 1 Day 1.
* Pregnant women are excluded from this study because ONC201 has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ONC201, breastfeeding should be discontinued if the mother is treated with ONC201. These potential risks may also apply to other agents used in this study.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ONC201.
* Patients who have known active Hepatitis B, or Hepatitis C infections.

INCLUSION CRITERIA FOR COHORT 2: TRIPLE NEGATIVE BREAST CANCER:

* Patients must have histologically or cytologically confirmed persistent or recurrent invasive, metastatic triple negative breast cancer (TNBC) for which standard curative measures do not exist or are no longer effective. TNBC, defined as estrogen receptor (ER) negative (ER < 10%), PR negative (PR <10%). HER2 will be considered negative per ASCO-CAP guidelines (HER2 test result as negative if a single test (or both tests) performed show: 1) IHC 1+ as defined by incomplete membrane staining that is faint/barely perceptible and within >10% of the invasive tumor cells; 2) IHC 0 as defined by no staining observed or membrane staining that is incomplete and is faint/barely perceptible and within less than or equal to 10% of the invasive tumor cells; or 3) ISH negative based on: a) Single-probe average HER2 copy number <4.0 signals/cell or b) Dual-probe HER2/CEP17 ratio <2.0 with an average HER2 copy number <4.0 signals/cell) and HER2 testing must have been performed in a laboratory accredited by the College of American Pathologists (CAP) or another accrediting entity.
* Patients must have received at least one line of prior chemotherapy in the metastatic setting.
* Patients must have measurable disease, per RECIST 1.1.
* Patients must have at least one lesion deemed safe to biopsy and be willing to undergo mandatory biopsies.
* Eligible patients may or may not have received prior chemotherapy and there is no limit to the number of prior chemotherapy. Patients are also eligible if they have received treatment with immunotherapy, such PD-1 inhibitors, PD-L1 inhibitors or cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) inhibitors.
* Age greater than or equal to 18 years.
* ECOG performance status 0 or 1
* Adequate renal function, defined as serum creatinine less than or equal to 1.5 X upper limit of normal (ULN), or measured creatinine clearance greater than or equal to 60 mL/min/1.
* Adequate hepatic function, defined as AST and ALT levels less than or equal to 3 X ULN and total bilirubin < 1.5 X ULN, unless known diagnosis of Gilbert's syndrome, where bilirubin less than or equal to 5 mg/dL will be permitted. Gilbert's syndrome will be defined as elevated unconjugated bilirubin, with conjugated (direct) bilirubin within the normal range and less than 20% of the total. Total bilirubin will be permitted up to 5 mg/dL, if patients have historical readings consistent with the definition of Gilbert's syndrome prior to entering study.
* Adequate bone marrow function, defined as absolute neutrophil (ANC) greater than or equal to 1,500/mm^3 (greater than or equal to 1.5 X10^6/L), platelet count greater than or equal to 75,000/mm^3 (greater than or equal to 75 X10^6/L), and hemoglobin greater than or equal to 9 mg/dL (transfusion to obtain hemoglobin greater than or equal to 9 mg/dL within 24 hours prior to dosing is allowed)
* Patients must be able to swallow oral medications (capsules) without chewing, breaking, crushing, opening or otherwise altering the product formulation.
* The effects of ONC201 on the developing human fetus are unknown. For this reason and because imipridone agents as well as other therapeutic agents used in this trial are known to be teratogenic. Female patients must either be of non-reproductive potential (i.e., post-menopausal by history: greater than or equal to 60 years old and no menses for greater than or equal to 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry and agree to use contraception or abstinence during the study and for and for at least 4 weeks after the final dose of any study-related medications. Male patients must use at least two forms of contraception during the study and for and for at least 4 weeks after the final dose of any study-related medications or have a partner who is not of reproductive potential.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA FOR COHORT 2: TRIPLE NEGATIVE BREAST CANCER:

* Patients who have received chemotherapy in the previous 3 weeks (6 weeks for nitrosoureas or mitomycin); other investigational agents within 3 weeks or a PD1/PDL1 agent within 4 weeks prior to first dose of study treatment.
* Patients who have undergone radiotherapy within 4 weeks of first dose of study treatment.
* Patients with a history of another invasive malignancy within the last 3 years.
* Patients with symptomatic brain metastases or leptomeningeal involvement. Patients with asymptomatic or brain metastases that have been treated with radiation at least 4 weeks prior to first dose of study treatment are allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to imipridones or other agents used in study.
* Patients with a mean QTcF interval of > 500 msec or receiving therapeutic agents known to prolong the QT interval
* Known history of cardiac arrhythmias including uncontrolled atrial fibrillation, tachyarrhythmias or bradycardia, history of congestive heart failure, or myocardial infarction or stroke in the previous 3 months will be excluded.
* Known history of gastrointestinal illnesses that would preclude the absorption of ONC201, which is an oral agent
* Patients with bone metastases who have initiated denosumab or bisphosphonate therapy within 28 days prior to Cycle 1 Day 1.
* Pregnant women are excluded from this study because ONC201 has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ONC201, breastfeeding should be discontinued if the mother is treated with ONC201. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ONC201.
* Patients who have known active Hepatitis B, or Hepatitis C infections.

INCLUSION CRITERIA FOR COHORT 3: ENDOMETRIAL CANCER:

* Patients must have histologically or cytologically confirmed persistent or recurrent advanced or metastatic invasive endometrial cancer (EC) for which standard curative measures do not exist or are no longer effective.
* Patients must have measurable disease, per RECIST 1.1
* Patients must have at least one lesion deemed safe to biopsy and be willing to undergo mandatory biopsies.
* Women with endometrial cancer must have had at least one prior line of therapy in the metastatic/recurrent setting but there is no limit to the number of prior chemotherapy lines. Patients are eligible if they have received treatment with immunotherapy, such PD-1 inhibitors, PD-L1 inhibitors or CTLA4 inhibitors.
* Age greater than or equal to 18 years.
* ECOG performance status 0 or 1
* Adequate renal function, defined as serum creatinine less than or equal to 1.5 X upper limit of normal (ULN), or measured creatinine clearance greater than or equal to 60 mL/min/1.
* Adequate hepatic function, defined as AST and ALT levels less than or equal to 3 X ULN and total bilirubin < 1.5 X ULN, unless known diagnosis of Gilbert's syndrome, where bilirubin less than or equal to 5 mg/dl will be permitted. Gilbert's syndrome will be defined as elevated unconjugated bilirubin, with conjugated (direct) bilirubin within the normal range and less than 20% of the total. Total bilirubin will be permitted up to 5 mg/dL, if patients have historical readings consistent with...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Lipkowitz, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Background] Greer YE, Lipkowitz S. TIC10/ONC201: a bend in the road to clinical development. Oncoscience. 2015 Feb 20;2(2):75-6. doi: 10.18632/oncoscience.133. eCollection 2015. No abstract available. PMID 25859547
- [Background] Endo Greer Y, Lipkowitz S. ONC201: Stressing tumors to death. Sci Signal. 2016 Feb 16;9(415):fs1. doi: 10.1126/scisignal.aad7955. PMID 26884598
- [Background] Stein MN, Bertino JR, Kaufman HL, Mayer T, Moss R, Silk A, Chan N, Malhotra J, Rodriguez L, Aisner J, Aiken RD, Haffty BG, DiPaola RS, Saunders T, Zloza A, Damare S, Beckett Y, Yu B, Najmi S, Gabel C, Dickerson S, Zheng L, El-Deiry WS, Allen JE, Stogniew M, Oster W, Mehnert JM. First-in-Human Clinical Trial of Oral ONC201 in Patients with Refractory Solid Tumors. Clin Cancer Res. 2017 Aug 1;23(15):4163-4169. doi: 10.1158/1078-0432.CCR-16-2658. Epub 2017 Mar 22. PMID 28331050
- [Derived] Atkins SLP, Greer YE, Jenkins S, Gatti-Mays ME, Houston N, Lee S, Lee MJ, Rastogi S, Sato N, Burks C, Annunziata CM, Lee JM, Nagashima K, Trepel JB, Lipkowitz S, Zimmer AS. A Single-Arm, Open-Label Phase II Study of ONC201 in Recurrent/Refractory Metastatic Breast Cancer and Advanced Endometrial Carcinoma. Oncologist. 2023 Oct 3;28(10):919-e972. doi: 10.1093/oncolo/oyad164. PMID 37279797
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0034.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1-Hormone Receptor (HR) + Breast Cancer (Male and Female); Cohort 2-Triple Negative Breast Cancer (Male and Female); Cohort 3-Endometrial Cancer (Female Only): 625mg ONC201 by mouth every 7 days
Period: Overall Study
Arm/Group | Cohort 1-Hormone Receptor (HR) + Breast Cancer (Male and Female) | Cohort 2-Triple Negative Breast Cancer (Male and Female) | Cohort 3-Endometrial Cancer (Female Only)
Started | 10 | 6 | 14
Completed | 7 | 5 | 10
Not Completed | 3 | 1 | 4
Not completed — Ineligible | 3 | 1 | 3
Not completed — Participant declined to participate before treatment started | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1-Hormone Receptor (HR) + Breast Cancer (Male and Female) | Cohort 2-Triple Negative Breast Cancer (Male and Female) | Cohort 3-Endometrial Cancer (Female Only) | Total
Number analyzed (Participants) | 10 | 6 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 8 | 22
  >=65 years | 2 | 0 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.14 (6.25) | 53.88 (8.37) | 63.65 (8.99) | 60.53 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 14 | 30
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 8 | 5 | 13 | 26
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 3 | 2 | 6
  White | 8 | 2 | 11 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1 - Progression-free Survival (PFS)
Description: PFS in participants with refractory, metastatic hormone receptor positive breast cancer. PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Progression is at least a 20% increase in the sum of the diameters of target lesions. And the appearance of one or more new lesions.
Time Frame: Every 8 weeks, while on the Trial. Participants were followed for an average of 8-10 weeks (up to 16 weeks).
Population: 7/10 participants were analyzed because 3 participants were ineligible.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1-Hormone Receptor (HR) + Breast Cancer (Male and Female)
Number analyzed (Participants) | 7
Months | 1.9 [0.6 to 4]

2. Primary Outcome: Cohort 2 - Overall Response Rate (ORR) (Complete Response (CR) + Partial Response (PR) by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Overall response (Complete response (CR) + Partial Response (PR) of ONC201 in participants with metastatic triple negative breast cancer was measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions.
Time Frame: Every 8 weeks, while on the Trial. Participants were followed for an average of 8-10 weeks (up to 16 weeks).
Population: 5/6 participants were analyzed because 1 participant was ineligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2-Triple Negative Breast Cancer (Male and Female)
Number analyzed (Participants) | 5
Participants
  Complete Response | 0
  Partial Response | 0

3. Primary Outcome: Cohort 3 - Overall Response Rate (ORR) (Complete Response (CR) + Partial Response (PR) by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Overall response (Complete response (CR) + Partial Response (PR) of ONC201 in participants with advanced or metastatic endometrial cancer was measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions.
Time Frame: Every 8 weeks, while on the Trial. Participants were followed for an average of 8-10 weeks (up to 16 weeks).
Population: 10/14 participants were analyzed because 3 participants were ineligible, and 1 participant declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3-Endometrial Cancer (Female Only)
Number analyzed (Participants) | 10
Participants
  Complete Response | 0
  Partial Response | 0

4. Secondary Outcome: Number of Serious and Non-serious Adverse Events Grade ≥1 in Cohorts 1, 2, and 3
Description: Serious and non-serious adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, , Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 13 months and 28 days for cohort 1, 11 months and 12 days for cohort 2, and 34 months and 29 days for cohort 3.
Population: 7/10 participants were analyzed in cohort 1 because 3 participants were ineligible. 5/6 participants were analyzed in cohort 2 because 1 participant was ineligible. And 10/14 participants were analyzed in cohort 3 because 3 participants were ineligible, and 1 participant declined to participate before treatment started. Serious adverse events are denoted by an *.
Measure: Number; unit: Adverse events
Groups:
- Cohort 1 - Grade 1; Cohort 2 - Grade 1; Cohort 3 - Grade 1: Grade 1 is mild.
- Cohort 1 - Grade 2; Cohort 2 - Grade 2; Cohort 3 - Grade 2: Grade 2 is moderate.
- Cohort 1 - Grade 3; Cohort 2 - Grade 3; Cohort 3 - Grade 3: Grade 3 is severe.
- Cohort 1 - Grade 4; Cohort 2 - Grade 4; Cohort 3 - Grade 4: Grade 4 is life-threatening.
- Cohort 1 - Grade 5; Cohort 2 - Grade 5; Cohort 3 - Grade 5: Grade 5 is death related to adverse event.
Arm/Group | Cohort 1 - Grade 1 | Cohort 1 - Grade 2 | Cohort 1 - Grade 3 | Cohort 1 - Grade 4 | Cohort 1 - Grade 5 | Cohort 2 - Grade 1 | Cohort 2 - Grade 2 | Cohort 2 - Grade 3 | Cohort 2 - Grade 4 | Cohort 2 - Grade 5 | Cohort 3 - Grade 1 | Cohort 3 - Grade 2 | Cohort 3 - Grade 3 | Cohort 3 - Grade 4 | Cohort 3 - Grade 5
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 5 | 5 | 5 | 5 | 5 | 10 | 10 | 10 | 10 | 10
Adverse events
  Abdominal distension | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abdominal pain | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Abdominal pain | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  Alkaline phosphatase increased | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0
  Anemia | 2 | 0 | 0 | 0 | 0 | 1 | 5 | 3 | 0 | 0 | 2 | 2 | 0 | 0 | 0
  *Anemia | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anorexia | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Arthralgia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Ascites | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0
  *Atrial flutter | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Back pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood bilirubin increased | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Breast pain | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Breast pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Cardiac arrest | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Confusion | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Constipation | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cough | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Dehydration | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Dehydration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Diarrhea | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  *Diarrhea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Dizziness | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
  *Dysarthria | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dysgeusia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dyspepsia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dyspnea | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  *Dyspnea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema limbs | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Epistaxis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Facial pain | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fall | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Fall | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 0 | 0
  *Fatigue | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fever | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Fever | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Flu like symptoms | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Flushing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastroesophageal reflux disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Headache | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Hot flashes | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperhidrosis | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Hypotension | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Insomnia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Laryngeal hemorrhage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lethargy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphedema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocyte count decreased | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0
  Malaise | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Memory impairment | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mucosal infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Myalgia | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Nausea | 3 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  *Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Nervous system disorders - Other, specify | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-cardiac chest pain | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Pain | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Pain in extremity | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Paresthesia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  *Peripheral sensory neuropathy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pleural effusion | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  *Pleural effusion | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Proteinuria | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  *Pneumonitis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritus | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash maculo-papular | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Rhinorrhea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  *Sepsis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Sinus tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  *Sinus tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  *Stroke | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  *Thromboembolic event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  *Transient ischemic attacks | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Tremor | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Tumor hemorrhage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Upper respiratory infection | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urinary tract infection | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Urinary tract infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Vaginal discharge | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Vaginal hemorrhage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Vascular access complication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Vomiting | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  *Vomiting | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Weight loss | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Wheezing | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Cohort 1 - Overall Response Rate (Complete Response (CR) + Partial Response (PR) by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Overall response (Complete response (CR) + Partial Response (PR) of ONC201 in participants with refractory, metastatic hormone receptor positive breast cancer was measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions.
Time Frame: Every 8 weeks, while on the Trial. Participants were followed for an average of 8-10 weeks (up to 16 weeks).
Population: 7/10 participants were analyzed because 3 participants were ineligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1-Hormone Receptor (HR) + Breast Cancer (Male and Female)
Number analyzed (Participants) | 7
Participants
  Complete Response | 0
  Partial Response | 0

6. Secondary Outcome: Number of Participants in Cohorts 1, 2, and 3 With Clinical Benefit
Description: Clinical benefit is Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (i.e., at least a 20% increase in the sum of the diameters of target lesions).
Time Frame: Every 8 weeks, while on the Trial. Participants were followed for an average of 8-10 weeks (up to 16 weeks).
Population: 7/10 participants were analyzed in cohort 1 because 3 participants were ineligible. 5/6 participants were analyzed in cohort 2 because 1 participant was ineligible. And 10/14 participants were analyzed in cohort 3 because 3 participants were ineligible, and 1 participant declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1-Hormone Receptor (HR) + Breast Cancer (Male and Female) | Cohort 2-Triple Negative Breast Cancer (Male and Female) | Cohort 3-Endometrial Cancer (Female Only)
Number analyzed (Participants) | 7 | 5 | 10
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 1 | 1 | 2

7. Secondary Outcome: Cohorts 2 and 3 - Progression-free Survival (PFS)
Description: PFS in participants with triple negative breast cancer and endometrial cancer. PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Progression is at least a 20% increase in the sum of the diameters of target lesions. And the appearance of one or more new lesions.
Time Frame: Every 8 weeks, while on treatment, up to 3 months
Population: 5/6 participants were analyzed in cohort 2 because 1 participant was ineligible. And 10/14 participants were analyzed in cohort 3 because 3 participants were ineligible, and 1 participant declined to participate before treatment started.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 2-Triple Negative Breast Cancer (Male and Female) | Cohort 3-Endometrial Cancer (Female Only)
Number analyzed (Participants) | 5 | 10
Months | 1.2 [0.5 to 1.8] | 2 [0.6 to 3]

8. Other Pre Specified Outcome: Here is the Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1-Hormone Receptor (HR) + Breast Cancer (Male and Female) | Cohort 2-Triple Negative Breast Cancer (Male and Female) | Cohort 3-Endometrial Cancer (Female Only)
Number analyzed (Participants) | 7 | 5 | 10
Participants | 7 | 5 | 10

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 13 months and 28 days for cohort 1, 11 months and 12 days for cohort 2, and 34 months and 29 days for cohort 3.
Description: 7/10 participants were analyzed in cohort 1 because 3 participants were ineligible. 5/6 participants were analyzed in cohort 2 because 1 participant was ineligible. And 10/14 participants were analyzed in cohort 3 because 3 participants were ineligible, and 1 participant declined to participate before treatment started.
Arm/Group | Cohort 1-Hormone Receptor (HR) + Breast Cancer (Male and Female) | Cohort 2-Triple Negative Breast Cancer (Male and Female) | Cohort 3-Endometrial Cancer (Female Only)
All-Cause Mortality (participants affected / at risk) | 2/7 | 1/5 | 2/10
Serious Adverse Events (participants affected / at risk) | 4/7 | 3/5 | 5/10
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1-Hormone Receptor (HR) + Breast Cancer (Male and Female) (N=7) | Cohort 2-Triple Negative Breast Cancer (Male and Female) (N=5) | Cohort 3-Endometrial Cancer (Female Only) (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1-Hormone Receptor (HR) + Breast Cancer (Male and Female) (N=7) | Cohort 2-Triple Negative Breast Cancer (Male and Female) (N=5) | Cohort 3-Endometrial Cancer (Female Only) (N=10)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (2) | 3 (3)
Alkaline phosphatase increased (Investigations) | 2 (3) | 1 (3) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (9) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 1 (3) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (3) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 4 (5)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 6 (7)
Fever (General disorders) | 2 (3) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (5) | 1 (2) | 4 (6)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (3) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, Balance issues (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT03394027/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT03394027/ICF_001.pdf